CLINICAL TRIAL: NCT05369871
Title: Evaluation of a Closed-loop System for the Treatment of Type 2 Diabetes at Home (DT2_2)
Acronym: Close2target
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabeloop (Industry)
Collaborators: Icadom (Industry); AGIR à Dom (Other); University Hospital, Grenoble (Other); Centre Hospitalier Annecy Genevois (Other); Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RCB 2020-A03429-30
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus Type 2 - Insulin-Treated

STUDY DESIGN:
Intervention Model Description: This is a 13-week interventional, randomized, controlled, crossover, open-label, multicenter main study, followed by an optional, open-label, additional 4-week study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed-loop system followed by open-loop system (Experimental): An interventional cross-over study:
  * six weeks in closed-loop system with Accu-Chek Insight pump and continuous glucose monitoring (CGM) :consisting of 2 weeks of adaptation where data will not be collected + 4 weeks
  * followed by six weeks in open-loop system with usual pump and CGM : consisting of 2 weeks of adaptation where data will not be collected + 4 weeks ,
  Followed by an optional additional study: 4 weeks in closed-loop system.
  Interventions: Device: Closed-loop system; Device: Open-loop system
- Open-loop system followed by closed-loop system (Experimental): An interventional cross-over study:
  * six weeks in open-loop system with usual pump and CGM : consisting of 2 weeks of adaptation where data will not be collected + 4 weeks
  * followed by six weeks in closed-loop system with Accu-Chek Insight pump and CGM (including two weeks of adaptation) : consisting of 2 weeks of adaptation where data will not be collected + 4 weeks
  Followed by an optional additional study: 4 weeks in closed-loop system.
  Interventions: Device: Closed-loop system; Device: Open-loop system

INTERVENTIONS:
Device: Closed-loop system — Closed-loop system consisting of a terminal including the Diabeloop algorithm that is associated with the Dexcom G6 CGM and the Accu-Chek Insight insulin pump.
Device: Open-loop system — Open-loop system consisting of a terminal without the Diabeloop algorithm that is associated with the Dexcom G6 CGM and the usual insulin pump.

SUMMARY:
The objective of this clinical trial is to study the feasibility of using a closed loop and its impact on glycemic control, in patients with type 2 diabetes (T2D) treated with insulin pumps.

DETAILED DESCRIPTION:
T2D is a condition that combines insulin resistance and relative insulin deficiency. T2D naturally evolves into an increasingly marked insulin deficiency that leads to the need for pancreatic replacement, by administering insulin.

Type 1 diabetes (T1D) requires an integral and immediate substitution of pancreatic insulin secretion. Artificial intelligence, through a self-learning algorithm, enables the automation and personalization of insulin delivery. These devices, called "closed loops" bring a real benefit for the patients included in the studies, by improving the glycemic balance, by reducing the number of hypo- and hyperglycemias but also by reducing the mental load associated with the disease, improving their quality of life.

The objective of this clinical trial is to study the feasibility of using a closed loop and its impact on glycemic control, in patients with T2D treated with insulin pumps.

A 13-week interventional, randomized, controlled, crossover, open-label, multicenter main study, followed by an optional, open-label, additional 4-week study is proposed to patients.

Main objective: study of the impact of the closed loop for 6 weeks, compared to 6 weeks in an open loop, on glycemic balance (evaluated by the time in range 70-180 mg/dL).

Secondary objectives: study of the impact of the closed loop for 6 weeks, compared to 6 weeks in an open loop, on:

* glycemic balance (others parameters)
* daily physical activity
* quality of sleep
* satisfaction with diabetes treatment
* quality of life
* treatment safety

Evaluation of the satisfaction of the use (usability) of the system at the end of the closed loop period.

ELIGIBILITY:
Inclusion Criteria :

* Patient > 18 years old
* Patient with a weight < 150 kg
* Patient with type 2 diabetes (T2D) treated by insulin pump for at least 6 months
* Patient with stable pharmacological treatment of diabetes for at least 6 months
* Patient equipped with a CGM or Flash Glucose Meter (FGM)
* Patient diagnosed with T2D by a diabetologist
* Patient treated with a total daily dose of insulin < 160 U/24 h
* Patient with an HbA1c < 10%.
* Patient affiliated to the social security system or beneficiary of such a system
* Patient able to read and understand the procedure, and in a condition to express consent for the study protocol

No Inclusion Criteria:

* Patient with type 1 diabetes
* Patient receiving less than 8 units of insulin per day
* Patients suffering from a serious illness or undergoing treatment that may affect the physiology of diabetes, i.e., interactions with glucose and/or insulin that may interfere with the medical device (e.g., steroid treatment)
* Patient with severe uncorrected hearing and/or visual acuity problems
* Patient not wishing to use rapid-acting insulin analog 100 U/mL
* Patient who has undergone pancreatectomy or whose pancreas is severely impaired
* Patients with severe renal impairment (clearance < 30 mL/min)
* Patient with reduced sensation of hypoglycemia
* Patient with highly unstable diabetes
* Patient who received a pancreas or islet transplant
* Patient undergoing dialysis
* Critically ill patient
* Patient with neuropathy
* Patient with retinopathy
* Patient currently participating or having participated in the month prior to inclusion in another clinical interventional research study that may have an impact on the study, this impact is left to the discretion of the investigator
* Persons referred to in articles L1121-5 to L1121-8 of the CSP: pregnant women, parturients, nursing mothers, persons deprived of liberty by judicial or administrative decision, persons under legal protection
* Subject who would receive more than 4500 euros in compensation due to his or her participation in other research involving the human person in the 12 months preceding this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Glycemic control evaluation for the 12-week main study | Day 84
  Impact of 6 weeks of closed-loop compared to 6 weeks of open-loop on the glycemic balance (time spent in the target 70-180 mg/dL).
  The data used for the analysis are the last 4 weeks of each 6-week sequence.

SECONDARY OUTCOMES:
Daily glycemic variability evaluation for the 12-week main study | Day 84
  Impact of 6 weeks of closed-loop compared to 6 weeks of open-loop on the daily glycemic variability measured by the coefficient of variation The data used for the analysis are the last 4 weeks of each 6-week sequence.
Daily glycemic variability evaluation for the 12-week main study | Day 84
  Impact of 6 weeks of closed-loop compared to 6 weeks of open-loop on the daily glycemic variability measured by the standard deviation.
  The data used for the analysis are the last 4 weeks of each 6-week sequence.
Daily time spent in hypoglycemia evaluation for the 12-week main study | Day 84
  Impact of 6 weeks of closed-loop compared to 6 weeks of open-loop on the percentage of daily time spent in hypoglycemia.
  The data used for the analysis are the last 4 weeks of each 6-week sequence.
Daily time spent in hyperglycemia evaluation for the 12-week main study | Day 84
  Impact of 6 weeks of closed-loop compared to 6 weeks of open-loop on the percentage of daily time spent in hyperglycemia.
  The data used for the analysis are the last 4 weeks of each 6-week sequence.
Daily amount of insulin administered evaluation for the 12-week main study | Day 84
  Impact of 6 weeks of closed-loop compared to 6 weeks of open-loop on the average daily amount of insulin administered.
  The data used for the analysis are the last 4 weeks of each 6-week sequence.
Daily glucose management indicator (GMI) corresponding to the estimated HbA1c | Day 84
  Impact of 6 weeks of closed-loop compared to 6 weeks of open-loop on the Glucose management indicator (GMI) measurement using CGM data.
  The data used for the analysis are the last 4 weeks of each 6-week sequence.
Daily physical activity evaluation for the 12-week main study | Day 84
  Impact of 6 weeks of closed-loop compared to 6 weeks of open-loop on the daily physical activity, measured by actimetry for 7 days.
Sleep quality evaluation for the 12-week main study | Day 84
  Impact of 6 weeks of closed-loop compared to 6 weeks of open-loop on the sleep quality (duration and fragmentation), measured by actimetry for 7 days.
Diabetes treatment satisfaction evaluation for the 12-week main study | Days 42 and 84 (according to the randomized arm)
  Impact of 6 weeks of closed-loop compared to 6 weeks of open-loop on the diabetes treatment satisfaction, measured by the Diabetes Treatment Satisfaction Questionnaire (DTSQ).
  The DTSQ questionnaire is composed by a score which has a minimum of zero and a maximum of 36. The higher the score, the more satisfied the patient is with their treatment.
Quality of life questionnaire for the 12-week main study | Days 42 or 84 (according to the randomized arm)
  Impact of 6 weeks of closed-loop compared to 6 weeks of open-loop on the quality of life, measured by a questionnaire.
  This questionnaire is composed of 10 items. For each item, there are 3 possible answers: "less well than before"; "same as before"; "better than before". A score will be calculated from the 10 items by adding 1 point for each improvement answer allowing the calculation of a score varying between 0 and 10. A high score represents a better improvement in quality of life.
Incidence of Adverse events evaluation for the 12-week main study (safety and tolerability) | Day 84
  Impact of 6 weeks of closed-loop compared to 6 weeks of open-loop on the treatment safety, measured by the number of adverse events
System satisfaction questionnaire evaluation | Days 42 or 84 (according to the randomized arm)
  Evaluation of the closed loop system satisfaction by an usability questionnaire
  This questionnaire is composed of 5 sections. Section 1 evaluates satisfaction with the use of the medical device and will be evaluated through a score varying between 10 and 50. A high score means that satisfaction with the use of the device is high.
  Section 3 evaluates the ease of use of the device and will be evaluated through a score varying between 16 and 80. A high score means that the system is easy to use.
  Sections 2, 4 and 5 will not be scored and will only be subject to descriptive analysis.
Glycemic control evaluation for the 4-week additional study | Day 112
  Impact of 4 weeks of closed-loop without meal declaration compared to 4 weeks of closed-loop with meal declaration on the glycemic balance (time spent in the target 70-180 mg/dL).
Daily glycemic variability | Day 112
  Impact of 4 weeks of closed-loop without meal declaration compared to 4 weeks of closed-loop with meal declaration on the daily glycemic variability measured by the coefficient of variation
Daily glycemic variability | Day 112
  Impact of 4 weeks of closed-loop without meal declaration compared to 4 weeks of closed-loop with meal declaration on the daily glycemic variability measured by the standard deviation
Percentage of daily time spent in hypoglycemia | Day 112
  Impact of 4 weeks of closed-loop without meal declaration compared to 4 weeks of closed-loop with meal declaration on the daily time spent in hypoglycemia
Percentage of daily time spent in hyperglycemia | Day 112
  Impact of 4 weeks of closed-loop without meal declaration compared to 4 weeks of closed-loop with meal declaration on the daily time spent in hyperglycemia
Average daily amount of insulin administered | Day 112
  Impact of 4 weeks of closed-loop without meal declaration compared to 4 weeks of closed-loop with meal declaration on the average daily amount of insulin administered
Daily glucose management indicator (GMI) corresponding to the estimated HbA1c | Day 112
  Impact of 4 weeks of closed-loop without meal declaration compared to 4 weeks of closed-loop with meal declaration on the Glucose management indicator (GMI) measurement using CGM data.
Diabetes treatment satisfaction | Day 112
  Impact of 4 weeks of closed-loop without meal declaration compared to 4 weeks of closed-loop with meal declaration on the diabetes treatment satisfaction, measured by the Diabetes Treatment Satisfaction Questionnaire.
  The DTSQ questionnaire is composed by a score which has a minimum of zero and a maximum of 36. The higher the score, the more satisfied the patient is with their treatment.
System satisfaction questionnaire evaluation | Day 112
  Evaluation of the system satisfaction by an usability questionnaire
  This questionnaire is composed of 5 sections. Section 1 evaluates satisfaction with the use of the medical device and will be evaluated through a score varying between 10 and 50. A high score means that satisfaction with the use of the device is high.
  Section 3 evaluates the ease of use of the device and will be evaluated through a score varying between 16 and 80. A high score means that the system is easy to use.
  Sections 2, 4 and 5 will not be scored and will only be subject to descriptive analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure BOREL, MD, PhD, Principal Investigator — CHU Grenoble Alpes
Locations (3):
- France (3):
  - CH Métropole Savoie, Chambéry
  - CH Annecy-Genevois, Epagny Metz-Tessy
  - CHU Grenoble Alpes, La Tronche

IPD SHARING:
Plan to Share IPD: No